CLINICAL TRIAL: NCT05716178
Title: Effectiveness of Trained Religious Leaders' Engagement in Maternal Health Education on Improving Maternal Health Service Utilization: Cluster Randomized Controlled Trial in Hadiya Zone, Southern Ethiopia
Brief Title: Effectiveness of Trained Religious Leaders' Engagement in Maternal Health Education in Ethiopia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jimma University (Other)
Collaborators: Wachemo University (Other)
Responsible Party: Principal Investigator, Abinet Arega Sadore, Assistant Professor, Jimma University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: RP0133/12
Record Dates: First submitted 2023-01-21; First posted 2023-02-08 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Maternal Health

STUDY DESIGN:
Intervention Model Description: The study will have two arms, i.e., intervention and control groups. The intervention group is assigned to receive training from religious leaders on maternal and neonatal health and the control group will be left to continue the routine practices.
Who Masked: Outcomes Assessor
Masking Description: The intervention will be single-blinded. The outcome assessors will be masked.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Maternal health education (Experimental): participants in the intervention group will receive behavioral change communication on maternal health from trained religious leaders. The local religious leaders from each clustered kebele will be recruited based on religious educational status (educational status greater than or equal to diploma), acceptance by their followers and popularity, in collaboration with religious organization leaders, health extension workers, and kebele leaders. Then after the potential religious leaders are recruited, the two days training will be given for them. Recruited religious leaders are expected to give training on the topics (maternal health) for four sessions to promote healthy maternal behaviors for the members of their religion. After training sessions, every participant will receive a copy of the visual materials (posters) containing the key messages for promoting prenatal health behaviors.
  Interventions: Behavioral: Maternal health education
- Usual or routine care (No Intervention): The control group in this study will be on the existing routine maternal service without a provision of religious leaders' training intervention. In this arm, there will be no intervention by the researchers, rather baseline and end line data will be collected.

INTERVENTIONS:
Behavioral: Maternal health education — The local religious leaders from each clustered kebele will be recruited based on religious educational status (educational status greater than or equal to diploma), acceptance by their followers and popularity, in collaboration with religious organization leaders, health extension workers, and kebele leaders. Then after the potential religious leaders are recruited, the two days training will be given for them. Recruited religious leaders are expected to give training on the topics (maternal health) for four sessions to promote healthy maternal behaviors for the members of their religion.
  Arms: Maternal health education

SUMMARY:
Community education and demand generation activities by involving family members, traditional and religious leaders in maternal health behaviours are potential solutions. Knowledge about maternal and neonatal health service utilization can be increased through community-based structures, such as religious organizations.

DETAILED DESCRIPTION:
Religious and faith community health promotions have the ability to reduce health inequities, and religious institutions are among the most respected and trustworthy institutions that can considerably boost public health work. Similarly, Faith leaders, in addition to physicians and health care providers, are another category of people who have a big impact on other people's beliefs, feelings, and behaviors, according to research. Spiritual leaders have the ability to impact health behavior on a variety of levels, from personal to ecological, with "knock-on" implications on community health. This is achieved via health education and health promoting strategies. Furthermore, the influence of faith leaders on health behavior is in line with the tenets of the Ottawa Charter for Health Promotion since they are perceived as strengthening community action. That is, communities must be empowered to participate in and govern their own affairs. A faith leader is in a unique position to encourage behavior change since he or she is a vital component of the community. According to an evaluation of programs involving faith-based organizations, clergy were able to considerably aid behaviour change, particularly among hard-to-reach populations. Other studies have also identified the importance of faith leader's influence on health behavior. Similarly, faith leaders influence on behavior has been attributed to Scripture-based passages that espouse the virtues of healthy living. Although some studies have suggested that spiritual leaders play a role in influencing congregants' health behaviors, little information on the amount of this influence and the mechanisms involved available.

In Ethiopia, the majority of the population belongs to a religious group, and religion is an important part of society. Through places of worship, religious institutions have access to a large portion of the population. Religious leaders serve as community leaders as well as gatekeepers of information and access to the population and can help raise awareness about underutilized maternal and neonatal health services. Therefore this cluster-randomized trial is designed to evaluate the effects of trained religious leaders' engagement in maternal health education in improving maternal health service utilization and knowledge of major obstetric danger signs.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women less than 20 weeks gestational age
* Living in selected kebele (small administrative unit in Ethiopia)
* Pregnant women willing to participate in the study

Exclusion Criteria:

• Pregnant women who are seriously ill and unable to communicate will be excluded from the study.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 612 (Estimated)
Dates: Start 2023-03 (Estimated); Primary Completion 2023-07 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Proportion of skilled delivery service utilization | one month
  Proportion of skilled delivery service utilization will be measured based on women who gave birth in health center and hospital by assistance of health professionals that have midwifery skills including Midwife nurse, Nurse, Health Officers and Doctors as reported by the participant.
Proportion of antenatal care service utilization | one month
  Proportion of antenatal care service utilization will be measured based on "at least one ANC attendance" (Women who have attended at least one ANC check-up during their current pregnancy) and "four or more ANC attendance" (Women who attended four or more ANC visits) during their current pregnancy as reported by the participant.

SECONDARY OUTCOMES:
Proportion of knowledge of major obstetric danger signs | one month
  Women who mention at least three neonatal danger signs will be considered to have good knowledge whereas those who mentioned less than three of the danger signs will be labelled to have poor knowledge as stated by several studies.
proportion of perception of pregnancy risk | one month
  It will be assessed by using self-report questionnaire consisting of 9 items designed to measure a pregnant woman's perception of her pregnancy risks. Each question has five options (1 = strongly disagree, 2 = disagree, 3 = neutral, 4 = agree, and 5 = strongly agree). Higher scores will indicate higher levels of perceived risk.
Proportion of birth preparedness and complication readiness | one month
  A woman will be classified as "well birth prepared" in the most recent pregnancy if she has accomplished three of the following practices: identified skilled health professional, saved money, identified transport or had delivery kit/materials. A woman who makes arrangements for birth in less than three of the four ways will be classified as "not well birth prepared".

CONTACTS AND LOCATIONS:
Overall Officials: Yohannes Kebede, PhD, Study Director — Jimma University
Locations (1):
- Hadiya Zone, Awasa, Southern Nations, Nationalities, and Peoples' Region, Ethiopia

IPD SHARING:
Plan to Share IPD: Yes
Baseline characteristics, outcome measure and statistical analysis
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Derived] Sadore AA, Kebede Y, Birhanu Z. Effectiveness of engaging religious leaders in maternal health education for improving maternal health service utilization in Ethiopia: cluster randomized controlled trial. Front Public Health. 2024 Jul 29;12:1399472. doi: 10.3389/fpubh.2024.1399472. eCollection 2024. PMID 39135926